CLINICAL TRIAL: NCT03683576
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled, Dose-ranging, Multi-center Study to Evaluate the Efficacy and Safety of GB001 as Maintenance Therapy in Adult Subjects With Moderate to Severe Asthma
Brief Title: GB001 in Adult Subjects With Moderate to Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GB001, Inc, a wholly owned subsidiary of Gossamer Bio, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gossamer Bio Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB001-2001
Record Dates: First submitted 2018-09-11; First posted 2018-09-25 (Actual); Results first posted 2021-08-23 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Asthma
Keywords: GB001; eosinophilic asthma; moderate asthma; severe asthma
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo once per day (QD) for 24 weeks
  Interventions: Drug: Placebo
- GB001 20 mg (Experimental): GB001 20 mg QD for 24 weeks
  Interventions: Drug: GB001
- GB001 40 mg (Experimental): GB001 40 mg QD for 24 weeks
  Interventions: Drug: GB001
- GB001 60 mg (Experimental): GB001 60 mg QD for 24 weeks
  Interventions: Drug: GB001

INTERVENTIONS:
Drug: GB001 — film-coated oral tablet
  Arms: GB001 20 mg; GB001 40 mg; GB001 60 mg
Drug: Placebo — film-coated oral tablet
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, dose-ranging, multi-center study to evaluate the efficacy and safety of GB001 when added to standard-of care (SOC) asthma maintenance therapy in adults with moderate to severe asthma and an eosinophilic phenotype with respect to asthma worsening at the end of 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria

* A diagnosis of asthma by a physician at least 12 months before Screening Visit.
* Treated with medium or high dose inhaled corticosteroid (ICS) plus additional controller for at least 12 months prior to Screening Visit. Subjects must maintain a stable ICS dose regimen during the 4 weeks prior to the Screening Visit.
* Forced Expiratory Volume in 1 second (FEV1) of ≤ 85% of predicted normal
* Demonstrated reversibility of at least 12% in FEV1
* Evidence of uncontrolled asthma
* Eosinophilic asthma
* No changes in ICS dose and compliant with standard of care asthma therapy during run-in period.

Exclusion Criteria

* Current smokers (any substance)
* Serious co-morbidities
* Fridericia's correction QT factor (QTcF) ≥450 msec (male) or ≥470 msec (female)
* Use of other investigational drugs within 30 days, or within 5 half-lives, whichever is longer, prior to Screening Visit
* Regular use of systemic corticosteroids or immunosuppressive treatments or monoclonal antibodies for asthma
* Pregnant or breastfeeding

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (116):
- United States (47):
  - Clinical Research Center of Albama, LLC, Birmingham, Alabama
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - California Allergy and Asthma Medical Group, Los Angeles, California
  - Southern California Institute for Respiratory Diseases, Inc., Los Angeles, California
  - North Bay Clinical Trials, Inc, Napa, California
  - Allergy, Asthma & Sinus Consultants, Inc, Riverside, California
  - Integrated Research of Inland, Inc., Riverside, California
  - Allergy & Asthma Medical Group and Research Center, A P.C., San Diego, California
  - Allergy and Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - Bensch Clinical Research LLC, Stockton, California
  - Pulmonary Associates, Colorado Springs, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Central Florida Pulmonary Group, PA, Altamonte Springs, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Emerald Coast Research Associates, Panama City, Florida
  - Allergy and Asthma Diagnostic Treatment Center, Tallahassee, Florida
  - Clinical Research Trials of Florida, Inc., Tampa, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Atlanta Allergy & Asthma Clinic, PA,, Marietta, Georgia
  - Atlanta Allergy & Asthma Clinic, PA, Stockbridge, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Allergy & Asthma Specialists, PSC, Owensboro, Kentucky
  - John Hopkins Asthma and Allergy Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Medicine, Ann Arbor, Michigan
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - American Health Research, Charlotte, North Carolina
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oklahoma Institute of Allergy & Asthma Clinical Research, LLC, Oklahoma City, Oklahoma
  - Crisor, LLC, Medford, Oregon
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Berks Schuylkill Respiratory Specialists, Ltd., Wyomissing, Pennsylvania
  - AAPRI Clinical Research Institute, Warwick, Rhode Island
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Corsicana Medical Research, LLC, Corsicana, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas
  - Allergy and Asthma Research Center, PA, San Antonio, Texas
  - Pulmonary Research of Abingdon, LLC, Abingdon, Virginia
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
  - University of Wisconsin School of Medicine and Public Health Asthma, Allergy, and Pulmonary Clinical Research, Madison, Wisconsin
- Austria (3):
  - Ordination Dr. Robert Voves, Feldbach
  - SALK University Hospital Salzburg, State Hospital Salzburg, Salzburg
  - Medical University of Vienna, Department of Internal Medicine II, Clinical Division of Pulmonolog, Vienna
- Belgium (4):
  - UCL Saint-Luc - Pneumology Department, Brussels
  - Pneumocare sprl, Erpent
  - UZ Gent - Department of Respiratory Medicine, Ghent
  - CHU de Charleroi - Site André Vésale, Montigny-le-Tilleul
- Canada (8):
  - Inspiration Research Limited, Toronto, Ontario
  - CHUM - Departement de pneumologie, Montreal, Quebec
  - Allergiste & Immunologue - Clinic/Outpatient Facility, Montreal, Quebec
  - Centre integre universitaire de sante et de services sociaux du Nord-de-I'lle-de-Montreal - Hopital du Sacre-Coeur de Montreal, Montreal
  - Dr. Jamie Del Carpio's Clinic, Montreal
  - Inspirational Research Limited, Toronto
  - C. I. C Mauricie Inc., Trois-Rivières
  - The Lung Centre, Vancouver General Hospital, Vancouver
- Czechia (9):
  - St. Anne's University Hospital Brno, Institute of Clinical Immunology and Allergology, Brno
  - University Hospital Hradec Kralove, Institute of Clinical Immunology and Allergollogy, Hradec Králové
  - MediTrial s.r.o., Jindřichův Hradec
  - PNEUMO-KV s.r.o., Karlovy Vary
  - Pulmonary Outpatient Clinic - Dr. Otakar Hokynar, Kralupy nad Vltavou
  - University Hospital Olomouc, Department of Allergology and Clinical Immunology, Olomouc
  - Medicon a.s., Prague
  - Pulmonary Outpatient Clinic Rokycany s.r.o., Rokycany
  - Outpatient Allergology and Neurology Clinic Kasmed Ltd., Tábor
- France (4):
  - La Croix Rousse Hospital, Lyon
  - Nord G&R Laennec Hospital, Nantes
  - Centre Hospitalier Annecy Genevois, Pringy
  - NOUVEL HOPITAL CIVIL - New Civil Hospital, Strasbourg
- Germany (12):
  - Universitatsklinikum des Saarlandes, Klinik fur Innere Medizin V, Homburg, Saarland
  - RCMS Dr. Linhoff, Berlin
  - Pneumologisches Studienzentrum Margrafenstrasse, Berlin
  - Institut fuer Allergie - und Asthmaforschung, Berlin
  - Pneumologische Praxis am Schloss, Berlin
  - IKF Pneumologie GmbH & Co. KG, Frankfurt am Main
  - Pneumologicum im Suedstadtforum, Hanover
  - Schmid, Koblenz
  - BAG Prof. Hoheisel/Dr. A. Bonitz, Leipzig
  - Pneumologische Praxis PD Dr. med., Leipzig
  - KLB Gesundheitsforschung Luebeck GmbH, Lübeck
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz - Hospital, Mainz
- Poland (10):
  - Centrum Medycyny Oddechowej Mroz sp. j., Bialystok
  - Malopolskie Centrum Alergologii, Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej (NZOZ), Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1, Lodz
  - Ostrowieckie Centrum Medyczne, Ostrowiec Świętokrzyski
  - SPZOZ Proszowice, Proszowice
  - Gabinet Lekarski Zenon Bukowczan, Sucha Beskidzka
  - ALL-MED - Specjalistyczna Opieka Medyczna - Medyczny Instytut Badawczy Marek Jutel, Wroclaw
  - Centrum Medyczne Melita Medical, Wroclaw
  - NZOZ Lekarze Specjalisci, Wroclaw
- Spain (6):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Instituto de Ciencias Medicas, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Doctor Peset, Valencia
- Ukraine (8):
  - Public Institution: Dnipro Clinical Association of Urgent Medical Care under Dnipro City Council, Dnipro
  - Public Institution "City Clinical Hospital #4" under Dnipro City Council, Dnipro
  - Ivano-Frankivsk Central City Clinical Hospital, Ivano-Frankivsk
  - Public Non-Profit Enterprise: City Clinical Hospital #13 under Kharkiv City Council, Kharkiv
  - State Organization "National Institute of Phthisiology and Pulmonolgy named after F.G. Yanovsky NAMSU", Kyiv
  - Public Institution: City Clinical Hospital #6, Zaporizhia
  - Public Non-Profit Enterprise City Hospital #1 under Zaporizhia City Council, Zaporizhia
  - Public Enterprise "Hospital #1" under Zhytomyr City Council, Zhytomyr
- United Kingdom (5):
  - Birmingham Heartlands Hospital, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Glasgow Clinical Research Facility, Glasgow Royal Infirmary, Glasgow
  - Royal Liverpool University Hospital, Liverpool
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moss MH, Lugogo NL, Castro M, Hanania NA, Ludwig-Sengpiel A, Saralaya D, Dobek R, Ojanguren I, Vyshnyvetskyy I, Bruey JM, Osterhout R, Tompkins CA, Dittrich K, Raghupathi K, Ortega H; LEDA Investigators. Results of a Phase 2b Trial With GB001, a Prostaglandin D2 Receptor 2 Antagonist, in Moderate to Severe Eosinophilic Asthma. Chest. 2022 Aug;162(2):297-308. doi: 10.1016/j.chest.2022.02.038. Epub 2022 Mar 3. PMID 35248549
- [Derived] Ortega H, Fitzgerald M, Raghupathi K, Tompkins CA, Shen J, Dittrich K, Pattwell C, Singh D. A phase 2 study to evaluate the safety, efficacy and pharmacokinetics of DP2 antagonist GB001 and to explore biomarkers of airway inflammation in mild-to-moderate asthma. Clin Exp Allergy. 2020 Feb;50(2):189-197. doi: 10.1111/cea.13524. Epub 2019 Nov 26. PMID 31659803

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a run-in period, during which eligibility for randomization was determined. 731 participants entered the run-in period, 481 of whom were randomized.
Period: Overall Study
Arm/Group | Placebo | GB001 20 mg | GB001 40 mg | GB001 60 mg
Started (Randomized and treated. One participant randomized to GB001 40 mg was never treated and was therefore excluded from the Intent-to-Treat (ITT) and Safety Analysis Populations.) | 120 | 120 | 118 | 122
Completed | 114 | 116 | 106 | 114
Not Completed | 6 | 4 | 12 | 8
Not completed — Withdrawal by Subject | 2 | 0 | 8 | 3
Not completed — Adverse Event | 3 | 0 | 0 | 4
Not completed — Lack of Efficacy | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2 | 0
Not completed — Other, Not Specified | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population: all participants who were randomized and received at least 1 dose of study treatment
Groups:
- Placebo: Placebo QD for 24 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | GB001 20 mg | GB001 40 mg | GB001 60 mg | Total
Number analyzed (Participants) | 120 | 120 | 118 | 122 | 480
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (11.91) | 52.8 (11.81) | 52.9 (13.32) | 49.9 (14.37) | 51.8 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 86 | 74 | 72 | 308
  Male | 44 | 34 | 44 | 50 | 172
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 108 | 109 | 109 | 112 | 438
  Black or African American | 6 | 7 | 8 | 6 | 27
  Asian | 4 | 3 | 0 | 1 | 8
  Other, Not Specified | 1 | 1 | 1 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 107 | 113 | 112 | 116 | 448
  Hispanic or Latino | 11 | 2 | 5 | 5 | 23
  Unknown or Not Reported | 2 | 5 | 1 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Experience Worsening of Asthma by Week 24
Description: Proportion of participants who experience worsening of asthma by Week 24 as defined by at least 1 of the following:
  * On 2 consecutive days, morning (AM) peak expiratory flow (PEF) ≤ 75% of mean AM PEF measured over the last 7 days of the Run-in
  * Forced expiratory volume in 1 second (FEV1) < 80% of baseline
  * Increase in rescue medication use of ≥ 6 puffs/day on 2 consecutive days compared to mean use over the last 7 days of the Run-in
  * Increase in Asthma Control Questionnaire 5 (ACQ-5; see Outcome Measure 2 for description) score of ≥ 0.5 compared to baseline
  * The occurrence of a severe asthma exacerbation (asthma attack) defined as deterioration of asthma that leads to the use of systemic corticosteroids for at least 3 days, hospitalization, or an Emergency Department visit.
Time Frame: up to Week 24
Population: ITT Population: all participants who were randomized and received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Placebo | GB001 20 mg | GB001 40 mg | GB001 60 mg
Number analyzed (Participants) | 120 | 120 | 118 | 122
proportion of participants | 0.658 [0.570 to 0.737] | 0.567 [0.477 to 0.652] | 0.568 [0.478 to 0.654] | 0.557 [0.469 to 0.642]
Statistical Analysis 1: Comparison: Placebo vs GB001 20 mg; Test type: Superiority; p = 0.1425, Regression, Logistic; Odds Ratio (OR) = 0.674, 95% CI 2-sided [0.398 to 1.142] — GB001 20 mg vs. Placebo
Statistical Analysis 2: Comparison: Placebo vs GB001 40 mg; Test type: Superiority; p = 0.1482, Regression, Logistic; Odds Ratio (OR) = 0.677, 95% CI 2-sided [0.399 to 1.149] — GB001 40 mg vs. Placebo
Statistical Analysis 3: Comparison: Placebo vs GB001 60 mg; Test type: Superiority; p = 0.1086, Regression, Logistic; Odds Ratio (OR) = 0.651, 95% CI 2-sided [0.385 to 1.100] — GB001 60 mg vs. Placebo

2. Secondary Outcome: Change From Baseline to Week 24 in Asthma Control Questionnaire - 5 (ACQ-5) Score
Description: The ACQ-5 is a 5-item questionnaire which has been developed as a measure of the participant's asthma control that can be quickly and easily completed. The questions are designed to be self-completed by the participant. The 5 questions enquire about the frequency and/or severity of symptoms in the prior week (nocturnal awakening, activity limitation, shortness of breath, wheeze). The response options for each of these questions consists of a zero (no impairment/limitation) to 6 (total impairment/limitation) scale.
Time Frame: Baseline, Week 24
Population: ITT Population: all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | GB001 20 mg | GB001 40 mg | GB001 60 mg
Number analyzed (Participants) | 120 | 120 | 118 | 122
score on a scale | -0.89 [-1.05 to -0.73] | -1.04 [-1.20 to -0.89] | -1.04 [-1.20 to -0.88] | -1.08 [-1.24 to -0.92]
Statistical Analysis 1: Comparison: Placebo vs GB001 20 mg; Test type: Superiority; p = 0.1647, ANCOVA; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.36 to 0.06] — GB001 20 mg vs. Placebo
Statistical Analysis 2: Comparison: Placebo vs GB001 40 mg; Test type: Superiority; p = 0.1737, ANCOVA; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.37 to 0.07] — GB001 40 mg vs. Placebo
Statistical Analysis 3: Comparison: Placebo vs GB001 60 mg; Test type: Superiority; p = 0.0879, ANCOVA; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.40 to 0.03] — GB001 60 mg vs. Placebo

3. Secondary Outcome: Change From Baseline to Week 24 in Pre-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: Pre-albuterol/salbutamol morning FEV1 was measured using electronic spirometry.
Time Frame: Baseline, Week 24
Population: ITT Population: all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: liters (L)
Arm/Group | Placebo | GB001 20 mg | GB001 40 mg | GB001 60 mg
Number analyzed (Participants) | 120 | 120 | 118 | 122
liters (L) | 0.105 [0.027 to 0.182] | 0.121 [0.041 to 0.200] | 0.146 [0.064 to 0.227] | 0.180 [0.102 to 0.257]
Statistical Analysis 1: Comparison: Placebo vs GB001 20 mg; Test type: Superiority; p = 0.7718, ANCOVA; Mean Difference (Net) = 0.016, 95% CI 2-sided [-0.091 to 0.123] — GB001 20 mg vs. Placebo
Statistical Analysis 2: Comparison: Placebo vs GB001 40 mg; Test type: Superiority; p = 0.4562, ANCOVA; Mean Difference (Net) = 0.041, 95% CI 2-sided [-0.067 to 0.149] — GB001 40 mg vs. Placebo
Statistical Analysis 3: Comparison: Placebo vs GB001 60 mg; Test type: Superiority; p = 0.1631, ANCOVA; Mean Difference (Net) = 0.075, 95% CI 2-sided [-0.030 to 0.180] — GB001 60 mg vs. Placebo

4. Secondary Outcome: Time to First Asthma Worsening
Description: Time to first asthma worsening is defined as the time from the date of the first dose of study treatment to the first date that any of the components of asthma worsening endpoint is met. See Outcome Measure 1 for the definition of asthma worsening.
Time Frame: up to Week 24
Population: ITT Population: all participants who were randomized and received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | GB001 20 mg | GB001 40 mg | GB001 60 mg
Number analyzed (Participants) | 120 | 120 | 118 | 122
weeks | 10.57 [7.857 to 16.286] | 17.43 [12.143 to NA] — NA (Not Available) indicates the value is not estimable due to an insufficient number of observed events. | 17.57 [13.429 to 24.286] | 19.86 [14.857 to NA] — NA (Not Available) indicates the value is not estimable due to an insufficient number of observed events.
Statistical Analysis 1: Comparison: Placebo vs GB001 20 mg; Test type: Superiority; p = 0.0466, Regression, Cox; Hazard Ratio (HR) = 0.719, 95% CI 2-sided [0.519 to 0.995] — GB001 20 mg vs. Placebo
Statistical Analysis 2: Comparison: Placebo vs GB001 40 mg; Test type: Superiority; p = 0.1222, Regression, Cox; Hazard Ratio (HR) = 0.773, 95% CI 2-sided [0.558 to 1.071] — GB001 40 mg vs. Placebo
Statistical Analysis 3: Comparison: Placebo vs GB001 60 mg; Test type: Superiority; p = 0.0304, Regression, Cox; Hazard Ratio (HR) = 0.698, 95% CI 2-sided [0.505 to 0.967] — GB001 60 mg vs. Placebo

5. Secondary Outcome: Annualized Rate of Severe Asthma Exacerbations
Description: A severe asthma exacerbation is defined as deterioration of asthma that leads to the use of systemic corticosteroids for at least 3 days, hospitalization, or an Emergency Department visit.
Time Frame: up to Week 24
Population: ITT Population: all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: events/year
Arm/Group | Placebo | GB001 20 mg | GB001 40 mg | GB001 60 mg
Number analyzed (Participants) | 120 | 120 | 118 | 122
events/year | 0.933 [0.664 to 1.311] | 0.744 [0.517 to 1.070] | 0.698 [0.480 to 1.015] | 0.829 [0.585 to 1.174]
Statistical Analysis 1: Comparison: Placebo vs GB001 20 mg; Test type: Superiority; p = 0.3382, Negative binomial regression model; Rate ratio = 0.797, 95% CI 2-sided [0.501 to 1.268] — GB001 20 mg vs. Placebo
Statistical Analysis 2: Comparison: Placebo vs GB001 40 mg; Test type: Superiority; p = 0.2248, Negative binomial regression model; Rate ratio = 0.748, 95% CI 2-sided [0.469 to 1.195] — GB001 40 mg vs. Placebo
Statistical Analysis 3: Comparison: Placebo vs GB001 60 mg; Test type: Superiority; p = 0.6090, Negative binomial regression model; Rate ratio = 0.889, 95% CI 2-sided [0.565 to 1.397] — GB001 60 mg vs. Placebo

6. Secondary Outcome: Change From Baseline to Week 24 in Post-Bronchodilator FEV1
Description: Post-albuterol/salbutamol morning FEV1 was measured using electronic spirometry.
Time Frame: Baseline, Week 24
Population: ITT Population: all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: L
Arm/Group | Placebo | GB001 20 mg | GB001 40 mg | GB001 60 mg
Number analyzed (Participants) | 120 | 120 | 118 | 122
L | 0.012 [-0.064 to 0.088] | -0.011 [-0.088 to 0.066] | 0.047 [-0.037 to 0.131] | 0.091 [0.015 to 0.166]
Statistical Analysis 1: Comparison: Placebo vs GB001 20 mg; Test type: Superiority; p = 0.6645, ANCOVA; Mean Difference (Net) = -0.023, 95% CI 2-sided [-0.127 to 0.081] — GB001 20 mg vs. Placebo
Statistical Analysis 2: Comparison: Placebo vs GB001 40 mg; Test type: Superiority; p = 0.5288, ANCOVA; Mean Difference (Net) = 0.035, 95% CI 2-sided [-0.074 to 0.144] — GB001 40 mg vs. Placebo
Statistical Analysis 3: Comparison: Placebo vs GB001 60 mg; Test type: Superiority; p = 0.1362, ANCOVA; Mean Difference (Net) = 0.079, 95% CI 2-sided [-0.025 to 0.182] — GB001 60 mg vs. Placebo

7. Secondary Outcome: Change From Baseline to Week 24 in Morning Peak Expiratory Flow (AM PEF)
Description: AM PEF was measured by participants using an electronic diary.
Time Frame: Baseline, Week 24
Population: ITT Population: all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Placebo | GB001 20 mg | GB001 40 mg | GB001 60 mg
Number analyzed (Participants) | 120 | 120 | 118 | 122
L/min | 8.993 [-1.514 to 19.499] | 15.115 [4.779 to 25.451] | 22.941 [12.042 to 33.839] | 14.581 [4.140 to 25.021]
Statistical Analysis 1: Comparison: Placebo vs GB001 20 mg; Test type: Superiority; p = 0.3957, ANCOVA; Mean Difference (Net) = 6.122, 95% CI 2-sided [-8.007 to 20.251] — GB001 20 mg vs. Placebo
Statistical Analysis 2: Comparison: Placebo vs GB001 40 mg; Test type: Superiority; p = 0.0598, ANCOVA; Mean Difference (Net) = 13.948, 95% CI 2-sided [-0.578 to 28.474] — GB001 40 mg vs. Placebo
Statistical Analysis 3: Comparison: Placebo vs GB001 60 mg; Test type: Superiority; p = 0.4376, ANCOVA; Mean Difference (Net) = 5.588, 95% CI 2-sided [-8.522 to 19.698] — GB001 60 mg vs. Placebo

8. Secondary Outcome: Percentage of Participants With a Treatment-Emergent Adverse Event (AE)
Description: An adverse event (AE) is any untoward medical occurrence in a participant, whether or not considered related to study treatment. Abnormal laboratory test results or other safety assessments, including those that worsened from baseline, that were considered clinically significant in the medical and scientific judgment of the investigator were to be reported as AEs.
Time Frame: From first dose of study treatment through Week 28
Population: Safety Population: all participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | GB001 20 mg | GB001 40 mg | GB001 60 mg
Number analyzed (Participants) | 120 | 120 | 118 | 122
percentage of participants | 65.8 | 65.8 | 69.5 | 68.0

ADVERSE EVENTS:
Time Frame: From first dose of study treatment through Week 28
Arm/Group | Placebo | GB001 20 mg | GB001 40 mg | GB001 60 mg
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120 | 0/118 | 1/122
Serious Adverse Events (participants affected / at risk) | 9/120 | 5/120 | 5/118 | 7/122
Other Adverse Events (participants affected / at risk) | 45/120 | 53/120 | 59/118 | 55/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | GB001 20 mg (N=120) | GB001 40 mg (N=118) | GB001 60 mg (N=122)
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Mineral metabolism disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | GB001 20 mg (N=120) | GB001 40 mg (N=118) | GB001 60 mg (N=122)
Nasopharyngitis (Infections and infestations) | 19 | 23 | 29 | 17
Sinusitis (Infections and infestations) | 3 | 4 | 10 | 3
Upper respiratory tract infection (Infections and infestations) | 7 | 3 | 8 | 4
Rhinitis (Infections and infestations) | 6 | 1 | 2 | 7
Bronchitis (Infections and infestations) | 6 | 4 | 1 | 1
Headache (Nervous system disorders) | 11 | 14 | 14 | 13
Hypertension (Vascular disorders) | 2 | 3 | 6 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 8
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 4 | 13
Alanine aminotransferase increased (Investigations) | 1 | 2 | 3 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT03683576/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT03683576/SAP_001.pdf